CLINICAL TRIAL: NCT04595864
Title: Neo-adjuvant Transarterial Chemoinfusion (TAI) for Patients With Hepatocellular Carcinoma Beyond Milan/UCSF Criteria Who Underwent Liver Transplantation
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Beicheng Sun, Director, Hepatobiliary Surgery, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: v1.0 20101014
Record Dates: First submitted 2020-10-13; First posted 2020-10-22 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Hepatocellular Carcinoma; Liver Transplantation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): Transarterial chemoinfusion (TAI) with mFOLFOX6 (oxaliplatin, calcium folinate, and 5-FU)
  Interventions: Other: Transarterial chemoinfusion (TAI) with mFOLFOX6 (oxaliplatin, calcium folinate, and 5-FU)
- control group (No Intervention): no neo-adjuvant treatment before operation

INTERVENTIONS:
Other: Transarterial chemoinfusion (TAI) with mFOLFOX6 (oxaliplatin, calcium folinate, and 5-FU) — TAI
  Other Names: TAI
  Arms: treatment group

SUMMARY:
Hepatocellular carcinoma (HCC) is the second commonest cause of cancer death worldwide. Liver transplantation (LT) is the best curative treatment of HCC meeting Milan/UCSF criteria. Milan (solitary tumour <5cm, or up to 3 tumours, each <3cm) and University of California San Francisco (UCSF) criteria (solitary tumour ≤6.5cm, up to 3 tumours with none >4.5cm, and total tumour diameter ≤8cm) provide the benchmark requirements for LT, at which a 5-year survival of >70% and recurrence rate ranging from 5-15% can be achieved.

Recently, FOLFOX (Oxaliplatin and 5-fluorouracil) based hepatic artery infusion chemotherapy (HAIC) exhibited high response rate for advanced HCC. Neo-adjuvant TAI for the HCC patients with beyond criteria serving as a down-staging method for the advanced HCC to meet Milan/UCSF criteria，and qualify for LT.

This study is to compare the impact on survival of neo-adjuvant TAI for patients with beyond Milan/UCSF Criteria HCC who underwent LT.

ELIGIBILITY:
Inclusion Criteria:

1. older than 18 years old and younger than 75 years listed for liver transplant;
2. ECOG PS≤1;
3. Child-Pugh Stage A or B
4. Proven hepatocellular carcinoma according patological examination or EASL/AASLD diagnostic criteria;
5. Not previous treated for tumor;
6. The tumor was diagnosed beyond Milan criteria or University of San Francisco criteria for LT
7. No distant metastasis;
8. The lab test could meet:

   Neutrophil count≥2.0×109/L; Hemoglobin≥100g/L; Platelet count≥75×109/L; Serum albumin≥35g/L; Total bilirubin<2-times upper limit of normal; ALT<3-times upper limit of normal; AST<3-times upper limit of normal; Serum creatine<1.5-times upper limit of normal; PT≤upper limit of normal plus 4 seconds; INR≤2.2;
9. Sign up consent.

Exclusion Criteria:

1. Cannot tolerate TAI or LT;
2. Distant metastasis exits;
3. Known history of other malignancy;
4. Be allergic to related drugs;
5. Be treated before (interferon included);
6. Known history of HIV infection;
7. Known history of drug or alcohol abuse;
8. Have GI hemorrhage or cardiac/brain vascular events within 30 days;
9. Pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
OS | From date of randomization until the date of death from any cause, assessed up to 60 months
  From date of randomization until the date of death from any cause, assessed up to 60 months

SECONDARY OUTCOMES:
RFS | From date of randomization until the date of recurrence, assessed up to 60 months
  recurrence-free survival
recurrence rate | 1 year, 2 year, 3 year, 5 year after surgery
  recurrence rate
PFS | From date of randomization until the date of progression, assessed up to 60 months
  progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Beicheng Sun, PhD，MD, Study Chair — Nanjing University
Locations (1):
- Nanjing Drum tower hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No